CLINICAL TRIAL: NCT00767338
Title: A Prospective, Randomized, Study of Microsurgical Varicocelectomy Versus Observation in the Treatment of Male Partners With a Palpable Varicocele and an Abnormal Semen Analysis
Brief Title: Microsurgical Varicocelectomy Versus No Surgery in Men With a Palpable Varicocele and an Abnormal Semen Analysis
Acronym: VIA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The DSMB recommended stopping the study because of concerns about the dismal recruitment, the drain on network resources, and the need for a study redesign.
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Penn State University (Other); University of Colorado, Denver (Other); University of Michigan (Other); University of Pennsylvania (Other); University of Texas (Other); University of Vermont (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Heping Zhang, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMN-VIA; 5U10HD055925-02 (NIH); 5U10HD055936 (NIH)
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Pregnancy; Infertility
Keywords: Infertility; Pregnancy; Men; Palpable varicocele; Abnormal semen analysis; Intrauterine insemination; Microsurgical varicocelectomy
MeSH Terms: conditions — Infertility; Multiple Endocrine Neoplasia Type 1 | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- No surgery + IUI (Active Comparator): No microsurgical varicocelectomy plus up to four cycles each of alternating intrauterine insemination and timed intercourse starting with intrauterine insemination.
  Interventions: Behavioral: Timed intercourse; Procedure: Intrauterine insemination
- No Surgery + TI (Active Comparator): No microsurgical varicocelectomy plus up to four cycles each of alternating intrauterine insemination and timed intercourse starting with timed intercourse.
  Interventions: Behavioral: Timed intercourse; Procedure: Intrauterine insemination
- Surgery + IUI (Active Comparator): Microsurgical varicocelectomy plus up to four cycles each of alternating intrauterine insemination and timed intercourse starting with intrauterine insemination.
  Interventions: Behavioral: Timed intercourse; Procedure: Microsurgical varicocelectomy; Procedure: Intrauterine insemination
- Surgery + TI (Active Comparator): Microsurgical varicocelectomy plus up to four cycles each of alternating intrauterine insemination and timed intercourse starting with timed intercourse.
  Interventions: Behavioral: Timed intercourse; Procedure: Microsurgical varicocelectomy; Procedure: Intrauterine insemination

INTERVENTIONS:
Behavioral: Timed intercourse — Timed intercourse
  Other Names: TI
Procedure: Microsurgical varicocelectomy — Microsurgical varicocelectomy
  Other Names: Surgery
  Arms: Surgery + IUI; Surgery + TI
Procedure: Intrauterine insemination — Intrauterine insemination
  Other Names: IUI

SUMMARY:
The primary research hypothesis is that microsurgical varicocelectomy will result in an increase in live birth in infertile couples where the male partner has a palpable varicocele and an abnormal semen analysis in comparison to male partners who do not have microsurgical varicocelectomy.

The secondary hypotheses include:

1. To assess whether up to 4 cycles of intrauterine insemination confers any additional increase in live birth rates compared to timed intercourse;
2. To examine spousal pregnancy rate as the secondary outcome; and
3. To study the effect of varicocelectomy in men with infertility, an abnormal semen analysis, and a palpable varicocele on

   * Testicular semen analysis parameters;
   * Serological measures of FSH, LH, total and free testosterone and
   * Measures of quality of life and sexual function in both partners.

DETAILED DESCRIPTION:
Study Design

This will be a randomized controlled clinical trial to examine the effect of varicocelectomy in men with infertility, an abnormal semen analysis, and a palpable varicocele. This approach will allow us to compare (i) the effect of microsurgical varicocelectomy on live birth rates after up to four cycles of alternating intrauterine insemination and four cycles of timed intercourse over 8 months and (ii) the relative effectiveness of intrauterine insemination versus timed intercourse on live birth rates. Secondary analyses will explore the effect of the surgical intervention on pregnancy rates, semen analysis parameters, serological hormonal measures in the male subjects, and quality of life measures in both the male and female partners.

Treatment

Two hundred and thirty-two couples will be randomized to the two intervention groups (microsurgical varicocelectomy plus up to four cycles each of alternating intrauterine insemination and timed intercourse or no microsurgical varicocelectomy plus up to four cycles each of alternating intrauterine insemination and timed intercourse).

Timing

We anticipate that it will take 3 years to complete the study. Enrollment will begin in year 1 of the study. 34 couples will need to be recruited per site over the duration of the study to reach the enrollment goal of 232 couples. Participants will be enrolled in the study for one year, with the male partner undergoing periodic study assessments at two month intervals.

ELIGIBILITY:
Inclusion Criteria:

* 6 months of infertility (primary or secondary - randomization will be stratified to allow equal numbers of primary and secondary infertility couples in the treatment vs. observation group), male partner > 18 years of age and < 50 years of age
* Female partner > 18 years of age and <= 40 years of age - randomization will be stratified for two groups - female partner <35 and female partner >=35
* Evidence of a hysterosalpingogram or Saline Infusion Sonogram with one patent tube and regular ovulatory cycles as defined by the recruiting site >25 days and <35 days in duration in the female partner
* Evidence of a bilateral grade I or unilateral grade II-III varicocele on physical exam in the male partner
* Abnormal semen analysis as defined by WHO II criteria with a sperm count of >5 X106 /ml or the presence of abnormal strict morphology as defined by Kruger criteria.

Exclusion Criteria:

* The presence of retrograde ejaculation or uncorrectable ejaculatory dysfunction
* Decreased ovarian reserve in the female partner as evidence by a day #3 FSH > 12 mIU/ml

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Nanette Santoro, MD, Study Chair — Albert Einstein College of Medicine; Gregory M Christman, MD, Principal Investigator — University of Michigan; Dana A Ohl, MD, Principal Investigator — University of Michigan; Richard Legro, MD, Study Director — Pennsylvania State University College of Medicine; Robert Brzyski, MD, PhD, Study Director — The University of Texas Health Science Center at San Antonio; Peter Casson, MD, Study Director — University of Vermont; Michael Diamond, MD, Study Director — Wayne State University; Heping Zhang, PhD, Study Director — Yale University; Christos Coutifaris, MD, Study Director — University of Pennsylvania; William D Schlaff, MD, Study Director — University of Colorado Denver Health Science Center
Locations (9):
- United States (9):
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Trussell JC, Christman GM, Ohl DA, Legro RS, Krawetz SA, Snyder PJ, Patrizio P, Polotsky AJ, Diamond MP, Casson PR, Coutifaris C, Barnhart K, Brzyski RG, Schlaff WD, Meacham R, Shin D, Thomas T, Zhang M, Santoro N, Eisenberg E, Zhang H; Reproductive Medicine Network. Recruitment challenges of a multicenter randomized controlled varicocelectomy trial. Fertil Steril. 2011 Dec;96(6):1299-305. doi: 10.1016/j.fertnstert.2011.10.025. PMID 22130101

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Surgery + IUI | No Surgery + TI | Surgery + IUI | Surgery + TI
Started | 1 | 2 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Surgery + IUI | No Surgery + TI | Surgery + IUI | Surgery + TI | Total
Number analyzed (Participants) | 1 | 2 | 0 | 0 | 3
Age Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 1 | 2 |  |  | 3
  >=65 years | 0 | 0 |  |  | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30 (0) | 33 (1) |  |  | 32 (2)
Gender [Number; unit: participants]
  Female | 0 | 0 |  |  | 0
  Male | 1 | 2 |  |  | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Live Births After Eight Cycles of Infertility Treatment.
Time Frame: January 2009 to January 2012
Population: The participants analyzed correspond to the number of participants who completed the study. In two of the arms, the study was terminated before participants were randomized to those arms.
Measure: Number; unit: participants
Arm/Group | No Surgery + IUI | No Surgery + TI | Surgery + IUI | Surgery + TI
Number analyzed (Participants) | 1 | 2 | 0 | 0
participants | 0 | 0 |  |

ADVERSE EVENTS:
Arm/Group | No Surgery + IUI | No Surgery + TI | Surgery + IUI | Surgery + TI
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No